CLINICAL TRIAL: NCT05607589
Title: A Phase 1, First-in-human, Randomized, Double-blind, Placebo Controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DWP213388 After SAD and MAD in Healthy Adult Subjects
Brief Title: The Safety, Tolerability, PK, and PD of DWP213388 After SAD and MAD Administration in Healthy Adult Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawal of Clinical Trial due to Licensing Out
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP213388101
Record Dates: First submitted 2022-10-19; First posted 2022-11-07 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DWP213388 (Experimental): Each cohort, healthy subjects will be administered DWP213388 (6 subjects per each cohort) SAD Cohort 1: DWP213388 x mg QD Cohort 2: DWP213388 x mg QD Cohort 3: DWP213388 x mg QD Cohort 4: DWP213388 x mg QD Cohort 5: DWP213388 x mg QD
  MAD Cohort 6: DWP213388 x mg QD Cohort 7: DWP213388 x mg QD Cohort 8: DWP213388 x mg QD Cohort 9: DWP213388 x mg QD
  Interventions: Drug: DWP213388
- Placebo (Placebo Comparator): Each cohort, healthy subjects will be administered placebo (2 subjects per each cohort) SAD Cohort 1: Placebo QD Cohort 2: Placebo QD Cohort 3: Placebo QD Cohort 4: Placebo QD Cohort 5: Placebo QD
  MAD Cohort 6: Placebo QD Cohort 7: Placebo QD Cohort 8: Placebo QD Cohort 9: Placebo QD
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DWP213388 — immunosuppressant
  Arms: DWP213388
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Phase 1, First-in-human, Randomized, Double-blind, Placebo controlled Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of DWP213388 after Single and Multiple Ascending Oral Dose Administration in Healthy Adult Subjects

DETAILED DESCRIPTION:
DWP213388 will be administered to the study subjects, according to a randomized, double-blind, and placebo-controlled design. The administration will be a single or multiple oral doses for healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign an Institutional Review Board (IRB) approved informed consent form (ICF) on a voluntary basis and to voluntarily participate in the study, after being fully informed of and completely understanding this study, prior to any screening procedure being undertaken.
2. Healthy adult male or female subject, of any race, between 18 to 65 years of age, inclusive at time of signing the ICF and prior to study intervention administration.
3. Body mass index (BMI) between 18.0 and 34.9 kg/m2 at Screening.
4. Subject who is determined to be in good health based on the results of medical history, physical examinations, 12-lead ECG, vital signs, and clinical laboratory evaluations at Screening or Day -1 as assessed by the Investigator (or designee).

Exclusion Criteria:

1. Subject has significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).

   attacks
2. Subject has fasting blood glucose > 110 mg/dL (> 6.1 mmol/L) (confirmed with repeat testing if required) at Screening.
3. Subject has a history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee). Please note subjects with allergies which can be managed without treatment can be included based on the decision of the Investigator (or designee).
4. Subject has a history of stomach or intestinal surgery or resection, including cholecystectomy, that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-02-20 (Estimated); Study Completion 2024-03-08 (Estimated)

PRIMARY OUTCOMES:
TEAE | up to 7 days from the last dosing
  Incidence and severity
12-lead ECG | up to 7 days from the last dosing
  PR interval, QRS interval, RR interval, QT interval, and QTcF

SECONDARY OUTCOMES:
Cmax | up to 72 hours from the last dosing
  Drug concentration in Blood and urine
AUC | up to 72 hours from the last dosing
  Area under curve
CL/F | up to 72 hours from the last dosing
  Clearance

CONTACTS AND LOCATIONS:
Overall Officials: Goldwater Ronald, Principal Investigator — Parexel